CLINICAL TRIAL: NCT05380544
Title: Extracorporeal Shockwave Therapy for Diabetic Foot Ulcers: A Pilot 3-Arm Randomised Control Trial and Qualitative Study (SOLEFUL).
Brief Title: Extracorporeal Shockwave Therapy for Diabetic Foot Ulcers
Acronym: SOLEFUL1
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R2743; 301807 (Other Grant/Funding Number: NIHR); 311664 (Other: IRAS)
Record Dates: First submitted 2022-04-22; First posted 2022-05-19 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Diabetic Foot
MeSH Terms: conditions — Diabetic Foot | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Pilot RCT and Qualitative study
Who Masked: Participant, Outcomes Assessor
Masking Description: Use of sham therapy for participant. Blinded outcome assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham shockwave therapy (Sham Comparator): Sham shockwave therapy in standard ulcer care.
  Interventions: Device: Extracorporeal Shockwave Therapy
- Low dose shockwave therapy (Active Comparator): 100 shocks per cm2 plus standard ulcer care
  Interventions: Device: Extracorporeal Shockwave Therapy
- High dose shockwave therapy (Active Comparator): 500 shocks per cm2 plus standard ulcer care
  Interventions: Device: Extracorporeal Shockwave Therapy

INTERVENTIONS:
Device: Extracorporeal Shockwave Therapy — ESWT will be given at 0.1mJ/mm2, 5 pulses/second and penetration of 5mm. Each intervention will be delivered in 3x30minute sessions over 7 days.

SUMMARY:
Summary of the problem:

Diabetes has been described as the fastest growing health crisis of our time. It currently affects more than 4.5million people in the UK. The direct cost to the NHS is already over £1 billion per year. One of the commonest complications of diabetes are foot ulcers. Despite current best treatment, these ulcers can be very difficult to heal, often taking months to heal and some never do. Even after healing ulcers return in up to 60% of people. In England someone undergoes an amputation of part of their foot every 2 hours and every 4 hours someone loses their leg due to diabetic foot ulcers. People are rarely able to be as active as before. This seriously affects their work, finances and quality of life.

Research into improved treatments are a national priority. These treatments need to be safe, effective, tolerable for patients and value for money. Preliminary research has identified shockwave therapy as a promising new treatment in which high-power soundwaves (similar to ultrasound) are delivered to the ulcer. This may make ulcers heal faster. However, the effectiveness of shockwave therapy and the optimum dose is unknown.

The aim of the study:

1. To carry out a preliminary (pilot) trial comparing sham (not active) shockwaves, low number of shockwaves and high number of shockwaves on diabetic foot ulcer healing
2. To understand beliefs, concerns, ideas and experience of shockwave therapy amongst patients and clinicians
3. To investigate the cost effectiveness (value for money) of shockwave therapy

Methods

1. Pilot Trial: Ninety patients with DFU will be randomly assigned to one of three treatment groups:

1. High dose shockwave treatment
2. Low dose shockwave treatment
3. "Sham" shockwave treatment

Each treatment will be delivered in 3x30minute sessions in a 7-day period. Face-to-face follow up appointments will take place 1, 2, 3 and 6 months after treatment to measure ulcer healing and changes in quality-of-life.

Interviews Interviews to explore patient opinion of shockwave therapy, experience in taking part in the trial, reasons patients do not want to take part and clinician attitudes to shockwave therapy

DETAILED DESCRIPTION:
There is an urgent need for better treatments for diabetic foot ulcers. Despite current best treatment, diabetic foot ulcers can be very difficult to heal, often taking months to heal and some never do. Even after healing ulcers return in up to 60% of people. In England someone undergoes an amputation of part of their foot every 2 hours and every 4 hours someone loses their leg due to diabetic foot ulcers. People are rarely able to be as active as before. This seriously affects their work, finances and quality of life.

This research is going to look at a new therapy called Extracorporeal Shockwave Therapy. Extracorporeal shockwave therapy (high power soundwaves) is a non-invasive treatment that is delivered directly to the ulcer and may improve healing. However, the effectiveness of shockwave therapy and the optimum dose is unknown. We will investigate if shockwave therapy improves diabetic foot ulcer healing. To do this we will undertake a randomised controlled trial. The trial will randomly allocate people (who are eligible to take part and consent) into one of three groups: sham shockwave therapy, low dose shockwave therapy and high dose shockwave therapy. The patient will not know which group they are in. The researcher collecting wound data will not know which group the patient is in. This is to ensure we and the patient do not influence the results of the study. This is a rigorous way of comparing new treatments to existing ones.

The purpose of the pilot trial is to provide information to be able to repeat this trial again with a larger number of people. This pilot trial will help identify any problems and address any issues before the main trial starts. This minimises the risk of wasting money and people's time.

The aim of this study is to:

* Carry out a preliminary (pilot) trial comparing sham (not active) shockwave therapy, low number of shockwaves and high number of shockwaves on diabetes foot ulcers
* To understand beliefs, concerns, ideas and experience of shockwave therapy amongst patients and clinicians

The research has been co-designed by patients and their families with experience of diabetic foot ulcers.

Pilot Trial:

The aim of the pilot trial is to see whether we can recruit enough patients to the study, how many patients remain in the study and reasons why patients leave the trial. It will also test whether we are collecting the information (data) in the right way to answer the research question. This is to make sure that the main trial is successful. Ninety patients who have a diabetic foot ulcer will be randomly assigned to one of the three treatment groups:

* High dose shockwave therapy
* Low dose shockwave therapy
* 'Sham' shockwave therapy

Each treatment will be delivered in a 3x30minute sessions over a 7 day period. All patients will receive usual ulcer care. Face to face follow up appointments will be at 6 weeks, 12 weeks and 24 weeks after study entry to measure ulcer healing, changes in quality of life and health resource use.

Interviews: Patients who are eligible to take part in the trial will be invited to an interview, to explore their reasons for (or for not) taking part, experience undergoing shockwave therapy and thoughts about being in the trial. This is to identify aspects of the trial which patients considered positive/negative so improvements can be made to the main trial. It will also help to improve the main trial and ensure our research is inclusive. Informal interviews, lasting around 30minutes, will be undertaken to explore patient opinion of shockwave therapy, experience of taking part in the trial, reasons patients do not want to take part and clinician attitudes to shockwave therapy. 24 patients and 8 clinicians will be invited to take part.

ELIGIBILITY:
Inclusion Criteria:

* At least one unhealed diabetic foot ulcer below the level of the medial malleoli that has been present for more than 4 weeks
* Absolute toe pressure greater than or equal to 50mmHg or an Ankle Pressure Brachial Index (ABPI) equal to or greater than 0.7(24, 25)
* Capacity to consent to participate in the trial and given written informed consent
* Willing to be randomised to either sham, low-dose or high-dose ESWT
* Willing to consent to photography of the index DFU
* Willing to comply with the follow up schedule

Exclusion Criteria:

* Interdigital index ulcer. This is because the ESWT delivery paddle does not fit between digits.
* Currently on or planned treatment for osteomyelitis.
* Currently taking any therapeutic anticoagulation medications. This includes novel oral anticoagulants, therapeutic doses of heparin and vitamin-K antagonists. This is a contraindication to ESWT.
* Diagnosis of malignancy in the treatment area or haematological, disseminated or lymphatic malignancy. This is a contraindication to ESWT.
* All who are pregnant, trying to conceive or breastfeeding. This is a contraindication to ESWT.
* Active participants in other trials that may conflict with the study outcomes, for example any other wound care trials.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2032-05-01 (Estimated)

PRIMARY OUTCOMES:
Eligibility ratio and recruitment ratio | 19 months
  Number eligible patients/number patients screened / recruited
Adherence to treatment | 19 months
  Number participants who completed the treatment protocol/number participants in the trial.
Percentage of missing data at each follow up point | 24 weeks
  Number of missing data points over number of data points x100
Follow up rates | 6 weeks
  No. of participants who attended each follow-up appointments / no. of follow-up appointments .
Follow up rates | 12 weeks
  No. of participants who attended each follow-up appointments / no. of follow-up
Follow up rates | 24 weeks
  No. of participants who attended each follow-up appointments / no. of follow-up
Patient and clinician acceptability of the trial process and ESWT | 24 weeks
  Semi-structured in depth interviews

SECONDARY OUTCOMES:
Time to DFU healing | 24 weeks
  Time taken for ulcer to heal
Proportion of DFUs healed at 6 months | 24 weeks
  The number of ulcers healed / total no. of ulcers healed in the trial
Reduction in ulcer size at each study visit | 24 weeks
  % reduction in ulcer size
Quality of life questionnaires | 24 weeks
  EQ-5L
Quality of life questionnaires | 24 weeks
  DFUS
Quality of life questionnaires | 24 weeks
  WoundQol
Adverse events | 24 weeks
  Instance of amputation, infection, mortality, side effects, re-hospitalisation
Cost differences between ESWT and standard care alone | 24 weeks
  Incremental Cost Effectiveness Ratio
Validity, reliability and responsiveness of WoundQol in patients with a DFU | 24 weeks
  To test WoundQol-14 reliability of the questionnaire in patients with a diabetic foot ulcer, participants will be asked to complete the questionnaire 3 days before the next follow-up appointment. The WoundQol-14 questionnaire will be repeated at the follow-up appointment. We will also test the validity of using WoundQol-14 over the telephone in patients who struggle to read (for example, due to diabetic retinopathy
Validity, reliability and responsiveness of virtual follow-up for wound healing in research | 24 weeks
  To test the feasibility, validity, reliability and responsiveness of virtual follow-up participants will be asked to send a photograph of their ulcer or ulcer site (if healed) 3 days before their follow up appointment to virtually assess the wound. Photographs are anticipated to be taken on the participant's smartphone by either themselves, a family member, friend or the community healthcare professional at dressing changes.

CONTACTS AND LOCATIONS:
Overall Officials: Louise Hitchman, MBBSMRCSMSc, Principal Investigator — Hull York Medical School
Locations (1):
- Hull University Teaching Hospitals NHS Trust, Hull, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data on request.
Supporting Information: Study Protocol, ICF
Time Frame: Data shared dependent on request, following study completion.
Access Criteria: Formal written letter to the PI.

REFERENCES:
- [Derived] Hitchman L, Iglesias C, Russell D, Smith G, Twiddy M, Chetter IC. A Pilot Three Arm Randomised Controlled Trial and Qualitative Study of Extracorporeal Shockwave Therapy for Diabetic Foot Ulcer Healing (SOLEFUL): A Study Protocol. Int Wound J. 2025 Apr;22(4):e70176. doi: 10.1111/iwj.70176. PMID 40159429